CLINICAL TRIAL: NCT07067203
Title: Correlation Between The Effect Of Quadriceps And Hamstring Strength On Timed Up And Go Scores In Adults With Tarns - Tibial Amputation
Brief Title: The Relationship of Quadriceps and Hamstring Strength on Timed up and go Scores in Transtibial Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmeen Essam Mohamed Abdelhafez, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P.T.REC/012/004809
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Amputation; Transtibial Amputation - Unilateral; Quadriceps Muscle Strength; Hamstring Muscle Strength; Timed Up and Go
Keywords: Transtibial amputation; transtibial amputee; Timed up and go; Hamstring muscle strength; quadriceps muscle strength; Transtibial amputation - unilateral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with Unilateral Transtibial Amputation (Experimental): Participants in this arm are adults aged 50 years or older with a unilateral transtibial amputation resulting from peripheral vascular disease or diabetic complications. All participants will have a K-level classification of 3 or 4 and a BMI within the normal range (18.5-29.9).
  Each participant will undergo two primary assessments:
  1. Muscle Strength Measurement
  2. Timed Up and Go (TUG) Test
  Interventions: Device: Lafayette hand held dynamometer; Diagnostic Test: Timed up and Go test

INTERVENTIONS:
Device: Lafayette hand held dynamometer — Muscle Strength Measurement:
  The strength of the quadriceps (knee extensors) and hamstrings (knee flexors) of the amputated limb will be measured using a handheld digital dynamometer (Nicholas MMT, Lafayette Instruments). Measurements will be taken with the prosthesis in place. Quadriceps strength will be assessed in a supine position with the knee at 30° flexion, while hamstring strength will be assessed in a prone position with the knee at 20° flexion. Each participant will perform three maximal effort trials after a practice attempt. The highest value will be scaled to body mass for analysis.
Diagnostic Test: Timed up and Go test — Timed Up and Go (TUG) Test:
  Participants will complete a standardized 3-meter TUG assessment to evaluate functional mobility. The test will be broken down into five components: standing, walking, turning, returning, and sitting. After one practice run, two timed trials will be conducted, and the average of both will be used for analysis. All procedures will be conducted by trained physical therapists following a standardized protocol.

SUMMARY:
To investigate the correlation between the effect of quadriceps and hamstring strength on timed up and go scores in adults with tarns - tibial amputation

DETAILED DESCRIPTION:
Lower limb amputation (LLA) has a significant socioeconomic and psychological impact on both individuals and communities. Despite these effects, major lower limb amputations remain relatively common worldwide. The causes of amputation vary by region, with the majority being non-traumatic in nature-most commonly linked to conditions such as diabetes mellitus, peripheral vascular disease, and cancer.

Individuals with lower limb amputation often experience musculoskeletal limitations, including reduced strength in the residual limb, limited range of motion (particularly in prosthetic joints), and challenges with postural control. As a result, they face a higher risk of falls compared to their able-bodied peers.

There has been limited research over the past two decades examining the use of the Timed Up and Go (TUG) test in adults with LLA. Since muscle strength plays a critical role in functional mobility, assessing the biomechanical and muscular conditions of individuals with amputation is essential for restoring daily function.

Unilateral amputation causes biomechanical asymmetries, making it important to monitor strength development in both the residual and intact limbs during prosthetic rehabilitation. Strength assessments can support balance recovery, improve movement confidence, and enhance gait performance.

Study Aim This study aims to explore the relationship between quadriceps strength in the amputated limb and Timed Up and Go (TUG) scores in adults with unilateral lower limb amputation. It will also investigate the association between hamstring strength and TUG scores in the same population.

ELIGIBILITY:
Inclusion Criteria:

1. All participants age 50 years or older, with the reason for amputation either peripheral vascular disease or diabetic complications (Nadollek & Brauer, 2002).
2. Unilateral transtibial amputation only (Wood, 2022).
3. K-level (2 to 4) (Gailey et al., 2002).
4. Normal Body mass index ranged from 18.5 to 30.0 (Nuttall, 2015).

Exclusion Criteria:

1. Residual limb revision in the past six months (Wood, 2022).
2. Open wounds or sores on the residual limb limiting the ability to don/doff prosthesis (Wood, 2022).
3. Uncontrolled comorbidities such as cardiovascular disease, active cancer treatment, and uncontrolled Diabetes Mellitus (Wood, 2022).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Correlation between the effect of quadriceps and hamstring strength by using Lafayette hand held dynamometer on the average of timed up and go scores in adults with tarns - tibial amputation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy College Cairo University, Giza, Egypt